CLINICAL TRIAL: NCT03155399
Title: Proprioceptive Stimulation With Manual Bilateral Rhythmic Exercise in Post-stroke Patients (Stimolazione Propriocettiva Manuale Con Esercizio Ritmico Bilaterale in Pazienti Post Ictus - BAT)
Brief Title: Proprioceptive Stimulation With Manual Bilateral Rhythmic Exercise in Post-stroke Patients
Acronym: BAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transferred to another Institution
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Pawel Kiper, PhD, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocollo 2012.07 BAT v.1.2
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Neurorehabilitation; Proprioceptive Training; Bilateral Arm Training; Intracortical Inhibition
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessment was conducted by two physiotherapists not involved in providing the experimental treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive based training (PBT) (Experimental): The treatment will last one hour and will be divided as follows: 2 proprioceptive based stimulation sessions per 3 minutes for each movement, with a rest of 2 minutes between each session. Every patient will receive 15 treatments, 5 days a week, for 3 weeks.
  Interventions: Other: Proprioceptive based training (PBT)
- Conventional neuromotor treatment (CNT) (Other): The CNT group will be treated for one hour daily by means of a CNT programme. The treatment will last 3 weeks.
  Interventions: Other: Conventional neuromotor treatment (CNT).

INTERVENTIONS:
Other: Proprioceptive based training (PBT) — During the PBT patient will stay in supine position with the upper limbs positioned in symmetric posture. He/She will be asked to move both limbs with the same frequency performing bilateral flexion-extension of one of the upper limb districts according to the available free ROM of the target joint. The movement execution of the affected arm will be supported by the physiotherapist performing passive movement at the same rhythm, as the one executed with the unaffected side. Patient will be asked to focus the attention on the movement performed against gravity, which will be reinforced by a verbal command. Afterwards, the physiotherapist will fully support movement execution coherently with the patient's movement initialization. The active movement performed voluntarily by the patient with unaffected limb will be considered as the reference movement, that the physiotherapist has to emulate passively, by synchronization of passive movement executed in phase with the affected side.
  Arms: Proprioceptive based training (PBT)
Other: Conventional neuromotor treatment (CNT). — The patients randomized to the CNT group will be asked to perform exercises for postural control, exercises for hand pre-configuration, exercises for the stimulation of manipulation and functional skills, exercises for proximal-distal coordination. All the exercises will be performed with or without the assistance of a physiotherapist. The upper limb motricity will be trained with progressive complexity.
  Arms: Conventional neuromotor treatment (CNT)

SUMMARY:
The purpose of this study is to evaluate the effect of the repetitive proprioceptive bilateral stimulation for the early recovery of the voluntary muscle contraction in stroke patients.

DETAILED DESCRIPTION:
The central nervous system (CNS) has plastic properties allowing its adaptation through development. These properties are still maintained in the adult age and potentially activated in case of brain lesion. In the present study authors hypothesized that a significant recovery of voluntary muscle contraction in post stroke patients experiencing severe upper limb paresis can be obtained, when proprioceptive based stimulations are provided. The proprioceptive based training (PBT) aims to stimulate the emergence of voluntary contraction and to foster motor recovery. It is based on motor learning principles, such as the repetition of tasks with concurrent use of feedbacks. The proposed concept is based on the concurrent repetitions of movements performed with the non-affected limb and with the affected one, passively mobilized by physiotherapist in charge of guaranteeing the optimal kinematic execution.

ELIGIBILITY:
Inclusion Criteria:

1. time since stroke up to 6 months,
2. presence of the upper limb plegia (0 point according to the Medical Research Council scale),
3. passive range of motion (ROM) completely free,
4. absence of primary joint trauma of the wrist, elbow and shoulder,

Exclusion Criteria:

1. increased muscle tone (score higher than 1 point in modified Ashworth scale),
2. apraxia (De Renzi test < 62 points),
3. global sensory aphasia (clinical notes),
4. neglect (clinical notes),
5. cognitive impairments (Mini Mental State Examination test < 24 points) ,
6. severe sensitivity disorders ( < 1 point in items shoulder, elbow, wrist and thumb at the proprioceptive sensitivity section of the Fugl-Meyer scale),
7. stroke lesion located in the cerebellum (clinical notes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Medical Research Council scale (MRC) | Change from baseline of the MRC scale at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions). The following muscles will be considered: deltoid, biceps brachii, triceps brachii, flexor carpi radialis, flexor carpi ulnaris, extensor carpi radialis, extensor carpi ulnaris, flexor digitorum and extensor digitorum.
Dynamometer | Change from baseline of dynamometer at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions)

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity scale (FM UE) | Change from baseline of the FM UE scale at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions).
Functional Independence Measure scale (FIM) | Change from baseline of the FIM scale at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions)
Modified Ashworth Scale | Change from baseline of the Ashworth scale at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions).
surface Electromyography (sEMG) | Change from baseline of the MVC at the end of PBT (three weeks thereafter)
  Applied at the beginning and at the end of treatment (after 15 sessions) and aiming to record the maximal voluntary contraction (MVC). sEMG signal will be recorded online during the tasks in each modality with bipolar electrodes from the following muscles; long head of biceps brachii, short head of biceps brachii, long head of triceps brachii and lateral head of triceps brachii.

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Kiper, PhD, Principal Investigator — Fondazione Ospedale San Camillo IRCCS; Andrea Turolla, PhD, Study Director — Fondazione Ospedale San Camillo IRCCS; Michela Agostini, MSc, Study Chair — Fondazione Ospedale San Camillo IRCCS; Alfonc Baba, MSc, Study Chair — Fondazione Ospedale San Camillo IRCCS
Locations (1):
- Fondazione Ospedale San Camillo IRCCS, Venezia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiper P, Szczudlik A, Venneri A, Stozek J, Luque-Moreno C, Opara J, Baba A, Agostini M, Turolla A. Computational models and motor learning paradigms: Could they provide insights for neuroplasticity after stroke? An overview. J Neurol Sci. 2016 Oct 15;369:141-148. doi: 10.1016/j.jns.2016.08.019. Epub 2016 Aug 11. PMID 27653881
- [Result] Kiper P, Baba A, Agostini M, Turolla A. Proprioceptive Based Training for stroke recovery. Proposal of new treatment modality for rehabilitation of upper limb in neurological diseases. Arch Physiother. 2015 Aug 3;5:6. doi: 10.1186/s40945-015-0007-8. eCollection 2015. PMID 29340175